CLINICAL TRIAL: NCT02574299
Title: Characterization of Ascending and Descending Auditory Processing Involved in the Encoding of Speech Sounds in Adult and Children: Variability Related to Changes in Sensory Input or a Neurodevelopmental Disorder or Targeted Remediation
Brief Title: Characterization of Auditory Processing Involved in the Encoding of Speech Sounds
Acronym: PRODIPRICIDE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2013-796; ID-RCB (Other: 2013-A00626-39)
Record Dates: First submitted 2015-08-14; First posted 2015-10-12 (Estimated); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Language Impairment; Hearing Loss
Keywords: dyslexia; training; auditory rehabilitation; hearing loss; evoked potentials; dichotic; plasticity; noise
MeSH Terms: conditions — Language Disorders; Hearing Loss; Dyslexia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- 1: Normal hearing children without SLI, transversal group (No Intervention): Normal hearing children without Specific Language Impairment (SLI),Transversal group for test-retest measures
- 2: Normal hearing children without SLI, longitudinal group (No Intervention): Normal hearing children without Specific Language Impairment (SLI), longitudinal group without training
- 3: Normal hearing children with SLI, longitudinal group (Other): Normal hearing children with Specific Language Impairment (SLI), longitudinal group with training
  Interventions: Other: E-learning
- 4: Normal hearing adults without SLI, transversal group (No Intervention): Normal hearing adults without Specific Language Impairment (SLI), transversal group for test-retest measures
- 5: Normal hearing adults without SLI, longitudinal group (No Intervention): Normal hearing adults without Specific Language Impairment (SLI), longitudinal group without hearing aids (HA)
- 6: Hearing Impaired candidates for HA, longitudinal group (Other): Hearing Impaired adult candidates for hearing aids (HA), longitudinal group with hearing aids (HA)
  Interventions: Device: Hearing aids fitting

INTERVENTIONS:
Other: E-learning — Management of auditory processing disorders with serious game (E-learning)
  Arms: 3: Normal hearing children with SLI, longitudinal group
Device: Hearing aids fitting — Symmetrical hearing loss which are fitted with binaural hearing aids for the first time
  Arms: 6: Hearing Impaired candidates for HA, longitudinal group

SUMMARY:
The ability to encode the speech signal is determined by ascending and descending auditory processing. Difficulties in processing these speech signals are well described at the behavioral level in a specific language disorder. However, little is known about the underlying pathophysiological mechanisms. The assumption is that we should observe a degradation of the signal provided by the ear in the deaf subject while in case of specific language impairment it would be a phonemic disorder (possibly linked to a processing disorder auditory). The two population groups should therefore have different abnormalities of their central auditory process - which could be modified by the target remediation for each group.

ELIGIBILITY:
Inclusion Criteria:

For all subjects:

* native French speaker
* no medical treatment for behavior or neurological disorders
* normal or corrected vision
* right-handed
* normal otorhinolaryngology examination
* valid affiliation to social security
* no participation to another research study

For the normal-hearing subjects

* normal tonal hearing thresholds
* normal tympanometry

For the subjects without specific language impairment

* aged from 6 ro 40
* normal school attendance without scholastic retardation
* normal intellectual level
* normal for age reading skills
* no delayed speech (expression & production)

For the children with specific language impairment

* aged fom 8 to 18
* persistent specific literacy difficulties with reading levels at least 18 months behind that of their peers
* normal intellectual level

For the hearing impaired subjects

* age from 18 to 70
* first auditory rehabilitation
* bilateral and symmetric hearing loss (±10 dB) with hearing thresholds between 0 and 25 dB at 0.25 kilohertz, 0 and 35 dB at 0.5 kilohertz, 0 and 50 dB at 1 kilohertz, 25 and 70 dB at 2 kilohertz, 25 and 80 dB at 3 kilohertz, 30 and 80 dB at 4 kilohertz

Exclusion Criteria:

* non signed assent
* treatment for depression, epilepsy, Parkinson's or alzheimer's disease during more than 6 months
* physical health deficiency
* mental retardation
* neurological or psychiatric disease incompatible with testing procedure

For children

* known problem of hearing loss or chronic middle ear disease whic compromized the hearing status
* schooling in a foreign language
* foreign language spoken at home with both parents

Ages: 6 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-10-16; Primary Completion 2018-03-01 (Actual); Study Completion 2018-03-01 (Actual)

PRIMARY OUTCOMES:
Change from Baseline speech auditory brainstem and late responses (composite and objective measure) in response to syllables (behavioral measure) | Arms 2 and 3: Baseline and 5 weeks / Arms 5 and 6: Baseline and 6 months / Arms 1 and 4: Baseline
  Spectro-temporal analysis of speech auditory brainstem and late responses : The speech brainstem and cortical responses are simultaneously obtained in response of different selected syllables from a continuum (selected by using a phonemic identification test) which is presented throughout a behavioral categorical procedure

SECONDARY OUTCOMES:
Change from Baseline medial olivocochlear system (MOCS) functioning measured using the contralateral suppressive effect of transient evoked otoacoustic emissions (composite measure) | Arms 2 and 3: Baseline and 5 weeks / Arms 5 and 6: Baseline and 6 months / Arms 1 and 4: Baseline
  Measurement of the contralateral suppressive effect of transient evoked otoacoustic emissions (expressed as Equivalent Attenuation)
Change from Baseline dichotic skills measured using central auditory processing tests (composite measure) | Arms 2 and 3: Baseline and 5 weeks / Arms 5 and 6: Baseline and 6 months / Arms 1 and 4: Baseline
  Presentation of different speech material to both ears simultaneously
Change from Baseline speech-noise listening skills measured using logatomes tests (composite measure) | Arms 2 and 3: Baseline and 5 weeks / Arms 5 and 6: Baseline and 6 months / Arms 1 and 4: Baseline
  Presentation of disyllabic words in presence of increasing noise levels

CONTACTS AND LOCATIONS:
Locations (1):
- Sercive d'Audiologie et d'Exploration Orofaciales, Hôpital Edouard Herriot, Hospices Civils de Lyon, Lyon, France

REFERENCES:
- [Result] Reynard P, Veuillet E, Thai-Van H. Paradoxical and labile medial olivocochlear functioning as a potential marker of auditory processing disorder in a child with learning disabilities. Eur Ann Otorhinolaryngol Head Neck Dis. 2020 Sep;137(4):339-342. doi: 10.1016/j.anorl.2020.03.005. Epub 2020 Apr 1. PMID 32247718
- [Result] Bellier L, Bouchet P, Jeanvoine A, Valentin O, Thai-Van H, Caclin A. Topographic recordings of auditory evoked potentials to speech: subcortical and cortical responses. Psychophysiology. 2015 Apr;52(4):594-9. doi: 10.1111/psyp.12369. Epub 2014 Oct 20. PMID 25329609
- [Result] Bellier L, Veuillet E, Vesson JF, Bouchet P, Caclin A, Thai-Van H. Speech Auditory Brainstem Response through hearing aid stimulation. Hear Res. 2015 Jul;325:49-54. doi: 10.1016/j.heares.2015.03.004. Epub 2015 Mar 27. PMID 25828076